CLINICAL TRIAL: NCT04366700
Title: Evaluate the Effect of Graft and Membrane on Healing of Apicomarginal Defects: A Randomized Controlled Trial
Brief Title: Evaluate the Effect of Graft and Membrane on Healing of Apicomarginal Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dr Sakshi
Record Dates: First submitted 2020-04-20; First posted 2020-04-29 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Apicomarginal Defects
Keywords: apicomarginal defects; autograft; prf; collagen membrane
MeSH Terms: interventions — Transplantation, Autologous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bone replacement substitute and membrane (Active Comparator): periapical surgery will be done and defect will be filled with a mixture of autograft and prf and over the defect and denuded root surface collagen membrane will be placed before closure of flap
  Interventions: Procedure: Periapical surgery with autograft and collagen membrane
- membrane (Active Comparator): periapical surgery will be done and defect will be filled with blood clot and over the defect and denuded root surface collagen membrane will be placed before closure of flap
  Interventions: Procedure: Periapical surgery with collagen membrane

INTERVENTIONS:
Procedure: Periapical surgery with autograft and collagen membrane — periapical surgery will be done and the defects will be filled with a mixture of autograft and prf and will be covered with a collagen membrane
  Arms: Bone replacement substitute and membrane
Procedure: Periapical surgery with collagen membrane — periapical surgery will be done and the defects will be filled with blood clot and covered with a collagen membrane
  Arms: membrane

SUMMARY:
This study will compare the effect of guided tissue regeneration using a mixture of autograft and PRF covered with a collagen membrane as compared to the membrane alone in the healing of apicomarginal defects. Healing of the lesions will be compared 2 dimensionaly and 3 dimensionaly using CBCT.

DETAILED DESCRIPTION:
Patients with apicomarginal defects as per the inclusion criteria will be randomly divided into two groups -in test group 1 -the defects will be filled with a mixture of autograft(which will be obtained from the surrounding buccal cortical plate by using a trephine bur) and prf(will be prepared by Choukron's method) and the defects and denuded root surface will be covered with a collagen membrane and in test group 2 -the defects will be filled with a blood clot and over that the collagen membrane will be placed. Radiographic and clinical healing will be assessed after 12 months, 2D healing will be assessed by Rud and Molven criteria and 3D healing will be assessed by Modified Penn 3D criteria.The clinical parameters recorded including periodontal pocket depth (PD), clinical attachment level (CAL) and gingival margin position (GMP) and will be measured on buccal aspect of the interproximal space and mid buccal aspect of the involved teeth using Williams 'O' periodontal probe.Routine examination procedure will be used to evaluate any evidence of signs and/or symptoms.. The criteria for a successful outcome included the absence of clinical signs and/or symptoms and radiographic evidence of complete or incomplete healing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age 16 years to 55 years
* Periapical defects with periodontal communication.
* Apicomarginal defects with probing depth > 6mm on mid-buccal and interproximal surfaces

Exclusion criteria

* Presence of buccal bone on flap elevation.
* Fractured /perforated roots.
* smokers.
* pregnant females and lactating mothers

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
change from baseline in periapical radiolucency at 12 months | Baseline to 12 months
  2 blinded caliberated operators will score the periapical radiolucency at baseline and 12 months by following scoring
  scores for 2D healing
  Score1-Complete healing defined by re-establishment of the lamina dura Score 2- Incomplete healing (scar tissue) Score 3- Uncertain healing Score 4- Unsatisfactory healing
  scores for 3D healing Score1- Complete healing Score 2- Limited healing Score 3- Uncertain healing Score 4- Unsatisfactory healing

SECONDARY OUTCOMES:
Clinical success | Baseline to 12 months
  Clinical success will be assessed by absence of clinical signs and symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Science, Rohtak, Haryana, India